CLINICAL TRIAL: NCT04720469
Title: A Safety Pilot Clinical Trial of a Second Magnetic Resonance Guided Focused Ultrasound (MRgFUS) Thalamotomy for the Management of Medication-refractory Essential Tremor
Brief Title: A Second Magnetic Resonance Guided Focused Ultrasound Thalamotomy for Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3341
Record Dates: First submitted 2020-11-05; First posted 2021-01-22 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-03

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Single-arm, pre/post designl study
Masking Description: This study is open label. CRST rating will be performed by a trained neurologist who will be blinded to whether the CRST data were collected pre- or post- treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with bilateral essential tremor who have undergone one MRgFUS thalamotomy (Experimental): Patients with bilateral essential tremor who have undergone one MRgFUS thalamotomy
  Interventions: Device: MRgFUS thalamotomy

INTERVENTIONS:
Device: MRgFUS thalamotomy — Ablation of untreated thalamus using focused ultrasound to abate tremor.
  Other Names: ExAblate Neuro

SUMMARY:
This study will be a single-centre, prospective, single-arm, open-label, 12-week pilot trial assessing the safety and preliminary efficacy of a second MR-guided focused ultrasound (MRgFUS) thalamotomy on the naïve brain hemisphere after 48 weeks or more of the first MRgFUS thalamotomy in patients with medication-refractory ET.

This study will be conducted at the Focused Ultrasound Centre of Excellence at Sunnybrook Health Sciences Centre/University of Toronto.

DETAILED DESCRIPTION:
Patients who are medication-refractory for ET often require a surgical option to relieve symptoms of ET and improve quality of life. To-date, unilateral MRgFUS has been beneficial in providing patients with some of relief from tremor. However, tasks that require two hands remain a challenge for many patients. Historical risks of bilateral treatment have been an impediment to complete tremor relief. The introduction of MRI and current stereotactic methodologies has significantly reduced the probability of non-target tissue injury. In this study, a second MRgFUS thalamotomy will be performed in a cohort of patients who have already successfully undergone unilateral MRgFUS treatment. Tremor severity, speech, balance, gait, and cognition will be assessed during baseline and follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 22 years or older;
2. Subjects who are able and willing to give consent and able to attend all study visits and MRgFUS procedure, understanding the associated risks, benefits, and alternative treatments;
3. Diagnosis of ET as confirmed from clinical history and examination by a neurologist or neurosurgeon and unilateral MRgFUS thalamotomy at least 48 weeks prior;
4. On a stable dose of medication for tremor for at least 4 weeks;
5. Medication-refractory criterion: tremor refractory to adequate trials of at least two medications, one of which should be a first line therapy of either propranolol or primidone. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated;
6. Moderate-severe tremor severity criteria in the untreated hand: Despite medical treatment, untreated hand score of ≥2 points in the postural or intention component of the item 5 or 6 in the Part A of CRST, AND untreated hand score of ≥2 points in any one of the items 12-15 of the Part B of CRST;
7. Disability criterion: ≥2 points in any one of the Part C items 17-23 as measured by the CRST;
8. Able to communicate sensations during the MRgFUS treatment and to press the device STOP button.

Exclusion Criteria:

1. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc;
2. Women who are pregnant;
3. Gait subscore ≥2 points in the SARA scale;
4. Speech subscore ≥2 points in the SARA scale;
5. Patients with advanced kidney disease (with estimated glomerular filtration rate <30 mL/min/1.73m2) or on dialysis;
6. Patients with unstable cardiac status or severe hypertension including:

   1. Documented myocardial infarction within six months of enrollment
   2. Unstable angina on medication
   3. Unstable or worsening congestive heart failure
   4. Left ventricular ejection fraction below the lower limit of normal
   5. History of a hemodynamically unstable cardiac arrhythmia
   6. Cardiac pacemaker
   7. Severe hypertension (diastolic BP > 100 on medication);
7. Patients exhibiting any behaviour(s) or clinical assessment consistent with ethanol or substance abuse;
8. Patients with history of abnormal bleeding, hemorrhage, and/or coagulopathy defined as abnormal coagulation profile (platelet < 100,00/μl), PT (>14 sec) or PTT (>36 sec), and INR > 1.3;
9. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure;
10. Ischemic or hemorrhagic stroke within 6 months;
11. Patients with brain tumors;
12. Individuals who are not able or unwilling to tolerate the required prolonged stationary position during treatment (approximately 2-3 hours);
13. Patients who are currently participating in another clinical investigation with an active treatment arm;
14. Patients who have had deep brain stimulation (DBS) or a prior stereotactic ablation of the basal ganglia with GKRS or radiofrequency;
15. Patients who have been administered botulinum toxins into the arm for 5 months prior to baseline.
16. Evidence of clinically important movement disorder, such as chorea, dystonia, or parkinsonism. Anyone with the presence of parkinsonian features including bradykinesia, rigidity, or postural instability will be excluded. Subjects who exhibit only mild resting tremor but no other symptoms or signs of Parkinson's disease may be included.
17. Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema);
18. Untreated, uncontrolled sleep apnea;
19. Presence of any other neurodegenerative disease like multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease;
20. Mild cognitive impairment with impairment in the domain of language as determined by screening neuropsychological battery and judged by study neuropsychologist;
21. A known diagnosis of dementia of any cause;
22. Uncontrolled major psychiatric disorder or suicidal ideation. Patients with psychiatric disorders identified on initial screening can be treated for these conditions before MRgFUS treatment and enrolled if deemed psychiatrically stable for at least three months before study entry. Any presence of psychosis will be excluded;
23. Any illness that in the investigator's opinion preclude participation in this study;
24. Patients with a history of seizures within the past year.
25. Inability to generate a thermal thalamic lesion during the first MRgFUS procedure;
26. Poor tolerance to the first MRgFUS procedure;
27. Severe adverse event or moderate-severe adverse event related to the MRgFUS procedure or thalamotomy, such as clinically significant and permanent speech, language, sensory, motor or gait dysfunction.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Incidence at week 12 of new onset or significant worsening of: ataxic gait; speech impairment; cognitive impairment; contralateral weakness; patient-reported disabling sensory loss; Severe AEs related to the MRgFUS procedure. | 12 weeks
  This composite outcome will be measured by the Scale for the Assessment and Rating of Ataxia (SARA) scale, neuropsychology battery, neurological examination and AE reports.

SECONDARY OUTCOMES:
Change in the tremor score (Part A and B) from baseline to 12 weeks after MRgFUS thalamotomy, adjusted for baseline scores. | 12 weeks
  This CRST subscore will be measured on the treated side.
Change in QUEST global score and EQ-5D from baseline to 12 weeks after MRgFUS, adjusted for baseline scores. | 12 weeks
  QUEST (Quality of Life in Essential Tremor) is a disease-specific quality of life scale.

OTHER OUTCOMES:
Change in speech intelligibility and speaking rate from baseline to 12 weeks after MRgFUS thalamotomy, adjusted for baseline scores. | 12 weeks
  Speech intelligibility is measured as the percentage of intelligible words and speaking rate is measured as words per minute.
Change in the subscores of neuropsychological tests and self-reported questionnaires from baseline to 12 weeks after MRgFUS thalamotomy. | 12 weeks
  Alternative versions of the neuropsychological tests and self-reported questionnaires of cognitive function will be used in the baseline and week 12 visit to account for a learning effect.

CONTACTS AND LOCATIONS:
Overall Officials: Agessandro Abrahao, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be made available by request and approval of the Sunnybrook REB and study PI.

REFERENCES:
- See also: Sunnybrook Focused Ultrasound Centre of Excellence — https://sunnybrook.ca/research/content/?page=sri-centres-focused-ultrasound-home